CLINICAL TRIAL: NCT00975403
Title: Pathophysiological Mechanisms of Dyspnea and Activity-Limitation in Mild COPD
Brief Title: Pathophysiological Mechanisms of Dyspnea and Activity-limitation in Mild Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Lung Association (Industry)
Responsible Party: Principal Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: DSS15110
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: mild COPD; dyspnea; exercise; respiratory mechanics; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dead space breathing (Experimental)
  Interventions: Device: Dead space breathing
- Room air breathing (Sham Comparator)
  Interventions: Device: Room air breathing

INTERVENTIONS:
Device: Dead space breathing — Chemical loading by adding a deadspace (600ml) to the breathing circuit during a single cycle exercise test
  Arms: Dead space breathing
Device: Room air breathing — Sham comparator (vs deadspace) during a single cycle exercise test will entail breathing room air on the same circuit without the rebreathe valves
  Arms: Room air breathing

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a growing cause of death, disability and health care costs in Canada. Nevertheless, COPD remains largely under-diagnosed and under-treated, particularly in its early stages. Patients with mild COPD have variable respiratory symptoms and often go unrecognized by their caregivers. Recent studies indicate that even smokers with near normal breathing test results can have extensive small airway disease/dysfunction at rest, which becomes more pronounced during the stress of exercise thus leading to unpleasant breathing difficulty. This study seeks to better understand the nature and causes of breathing discomfort and activity limitation in a group of patients with mild COPD. The investigators will compare detailed tests of small airway function and conduct an evaluation of several key physiological parameters during the stress of exercise in patients with mild COPD and in healthy, age-matched, non-smoking control subjects. The investigators will also compare detailed physiological responses to exercise under conditions of chemical loading and mechanical unloading of the respiratory system in patients with mild COPD.

The proposed study will be the first to systematically test the hypothesis that pathophysiological abnormalities in ventilatory demand, pulmonary gas exchange, small airway function, dynamic ventilatory mechanics and respiratory muscle function contribute significantly to exertional dyspnea and activity-limitation in patients with mild COPD. This study will be the first to determine if these abnormalities can be manipulated.

ELIGIBILITY:
Inclusion Criteria:

* Post-bronchodilator forced expiratory volume in 1 sec (FEV1) ≥ 80%predicted and a FEV1/forced vital capacity (FVC) ratio < 0.70;
* Clinically stable as defined by no changes in medication dosage or frequency of administration with no exacerbations or hospitalizations in the preceding 6 weeks;
* A cigarette smoking history ≥ 20 pack-yrs;
* Body mass index between 18.5 and 30 kg/m2;
* Able to perform all study procedures and provide informed consent.

Exclusion Criteria:

* A diffusing capacity of the lung for carbon monoxide (DLCO) < 40 %predicted;
* Presence of active cardiopulmonary disease (or comorbidities) other than COPD that could contribute to dyspnea and exercise limitation;
* Clinical diagnosis of sleep disordered breathing;
* History or clinical evidence of asthma;
* Presence of important contraindications to clinical exercise testing, including inability to exercise because of neuromuscular or musculoskeletal disease(s);
* Use of daytime oxygen or exercise-induced arterial oxygen desaturation to <80% on room air.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Dyspnea intensity measured by the 10-point Borg scale during cycle exercise | Standardized time during exercise

SECONDARY OUTCOMES:
Cycle exercise endurance time | During exercise testing at study visits

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, FRCPC, Principal Investigator — Queen's University and Kingston General Hospital
Locations (1):
- Respiratory Investigation Unit, Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Chin RC, Guenette JA, Cheng S, Raghavan N, Amornputtisathaporn N, Cortes-Telles A, Webb KA, O'Donnell DE. Does the respiratory system limit exercise in mild chronic obstructive pulmonary disease? Am J Respir Crit Care Med. 2013 Jun 15;187(12):1315-23. doi: 10.1164/rccm.201211-1970OC. PMID 23590271